CLINICAL TRIAL: NCT04158739
Title: A Phase 1 Trial of the CD123 X CD3 DART Molecule Flotetuzumab (NSC#808294) in Children, Adolescents, and Young Adults With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Flotetuzumab for the Treatment of Pediatric Recurrent or Refractory Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEPN1812; NCI-2019-06780 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PEPN1812 (Other: Pediatric Early Phase Clinical Trial Network); PEPN1812 (Other: CTEP); UM1CA228823 (NIH)
Record Dates: First submitted 2019-10-15; First posted 2019-11-12 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cytarabine, flotetuzumab) (Experimental): Patients receive cytarabine IT on days -6 to 0 prior to cycle 1. Patients may receive additional doses of cytarabine on day 1 of subsequent cycles per physician discretion. Patients also receive flotetuzumab IV continuously for 28 days. Treatment repeats every 29 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Biological: Flotetuzumab

INTERVENTIONS:
Drug: Cytarabine — Given IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Biological: Flotetuzumab — Given IV
  Other Names: CD123 x CD3 DART Bi-Specific Antibody MGD006; CD123 x CD3 Dual Affinity Re-Targeting Bi-Specific Antibody MGD006; MGD006; RES234; S80880

SUMMARY:
This phase I trial studies the side effects, best dose of flotetuzumab and how well it works in treating patients with acute myeloid leukemia (AML) that has come back (recurrent) or has not responded to treatment (refractory). This study also determines the safest dose of flotetuzumab to use in children with AML. As an immunotherapy, flotetuzumab may also cause changes in the body's normal immune system, which are also under study in this trial.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of flotetuzumab administered by continuous intravenous (IV) infusion to pediatric patients < 21 years of age with relapsed or refractory acute myeloid leukemia (AML).

II. To estimate the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of flotetuzumab administered by continuous IV infusion to pediatric patients < 21 years of age with relapsed or refractory AML.

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetics of flotetuzumab in pediatric patients with relapsed or refractory AML.

II. To preliminarily define the anti-tumor activity of flotetuzumab within the confines of a phase 1 study and correlate potential activity with baseline disease burden at study entry.

III. To monitor anti-drug antibody (ADA) production and characterize the immunogenicity of flotetuzumab.

EXPLORATORY OBJECTIVES:

I. To evaluate changes in T-lymphocyte population numbers before and after flotetuzumab treatment.

II. To evaluate the tumor microenvironment and cytokine production by immune effector cells before and after flotetuzumab treatment.

III. To quantify CD123 surface expression on AML cells at baseline and evaluate expression as a potential biomarker of flotetuzumab response.

OUTLINE: This is a dose-escalation/dose de-escalation study of flotetuzumab.

Patients receive cytarabine intrathecally (IT) on days -6 to 0 prior to cycle 1. Patients may receive additional doses of cytarabine on day 1 of subsequent cycles per physician discretion. Patients also receive flotetuzumab IV continuously for 28 days. Treatment repeats every 29 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must weigh >/= 17 kg

  * Weight limit is due to constraints related to the concentration of the current drug formulation. If a new formulation of flotetuzumab becomes available to allow dosing of smaller patients, the protocol will be amended.
* Patients with recurrent or refractory AML are eligible. Patients must have histologic verification of malignancy at relapse.
* Patients with leukemia must have >/= M2 marrow by morphology and/or flow cytometry and one of the following:

  * Second or greater relapse
  * Refractory after 2 or more chemotherapy cycles
  * First relapse after primary chemotherapy-refractory disease
  * First relapse after hematopoietic stem cell transplantation (HSCT)
* Central nervous system (CNS) disease:

  * Patients must have the status of CNS1 and no clinical signs or neurologic symptoms suggestive of CNS leukemia, such as cranial palsy.
  * Patients with CNS3 or CNS2 status may receive antecedent intrathecal chemotherapy to achieve CNS1 status prior to study entry.
  * Patients with a history of CNS chloromatous disease are required to have no radiographic evidence of disease prior to enrollment.
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =/< 16 years of age. Use appropriate score for study population. NOTE: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met, e.g., blood count criteria, the patient is considered to have recovered adequately.

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive.

    * >/= 14 days must have elapsed after the completion of other cytotoxic therapy with the exception of hydroxyurea. Additionally, patients must have fully recovered from all acute toxic effects of prior therapy.

      * NOTE: Cytoreduction with hydroxyurea is recommended to be discontinued >/= 24 hours prior to the start of protocol therapy. No waiting period is required for patients having received intrathecal cytarabine, methotrexate, and/or hydrocortisone.
  * Anti-cancer agents not known to be myelosuppressive (e.g., not associated with reduced platelet or absolute neutrophil count [ANC] counts): >/= 7 days after the last dose of agent.
  * Antibodies: >/= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =/< 1.
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, >/= 14 days must have elapsed since last dose of corticosteroid.
  * Hematopoietic growth factors: >/= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair and the study-assigned research coordinator.
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >/= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors).
  * Stem cell infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or stem cell boost: >/= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Donor leukocyte infusion: >/= 42 days
    * Autologous stem cell infusion including boost infusion: >/= 42 days
  * Cellular therapy: >/= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >/= 14 days after local XRT; >/= 84 days after TBI, craniospinal XRT or if radiation to >/= 50% of the pelvis; >/= 42 days if other substantial bone marrow (BM) radiation
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I-MIBG): >/= 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have received prior exposure to flotetuzumab.
* Platelet count >/= 20,000/mm^3 (may receive platelet transfusions)

  * These patients must not be known to be refractory to red cell or platelet transfusion
* Hemoglobin >/= 8.0 g/dL at baseline (may receive red blood cell [RBC] transfusions)

  * These patients must not be known to be refractory to red cell or platelet transfusion.
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >/= 70 ml/min/1.73 m^2 or
* A serum creatinine based on age/gender as follows:

  * Age: Maximum serum creatinine (mg/dL)

    * 1 to < 2 years: male - 0.6; female - 0.6
    * 2 to < 6 years: male - 0.8; female - 0.8
    * 6 to < 10 years: male - 1; female - 1
    * 10 to < 13 years: male - 1.2; female - 1.2
    * 13 to < 16 years: male - 1.5; female - 1.4
    * >/= 16 years: male - 1.7; female - 1.4
* Bilirubin (sum of conjugated + unconjugated) =/< 1.5 x upper limit of normal (ULN) for age regardless of baseline
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =/< 3 x ULN. For the purpose of this study, the ULN for SGPT is 45 U/L regardless of baseline.
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST/< 3 x ULN. For the purpose of this study, the ULN for SGPT is 50 U/L regardless of baseline.
* Serum albumin >/= 2 g/dL
* Shortening fraction of >/= 27% by echocardiogram, or
* Ejection fraction of >/= 50% by gated radionuclide study
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
* Nervous system disorders (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5) resulting from prior therapy must be =/< grade 2 with the exception of decreased tendon reflex (DTR). Any grade of DTR is eligible.
* All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
* Permanent central access should be established with a central line. A central line that contains 2 lumens is preferred.

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study because there is yet no available information regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of study therapy and for 12 weeks after flotetuzumab discontinuation.
* Patients must be off steroids (unless physiologic replacement dosing) for at least 7 days prior to enrollment. If used to modify immune adverse events related to prior therapy, >/= 14 days must have elapsed since last dose of corticosteroid.
* Patients who are currently receiving another investigational drug are not eligible.
* Patients who are currently receiving other anti-cancer agents are not eligible (except hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy).
* Patients who are receiving cyclosporine, tacrolimus or other agents to treat graft-versus-host disease post bone marrow transplant are not eligible for this trial.
* Patient has French-American-British classification (FAB) type M3 leukemia (acute promyelocytic leukemia) or identification of t(15;17).
* Patient has isolated CNS involvement or isolated extramedullary relapse.
* Patient with known human immunodeficiency virus (HIV) infection are eligible if he or she has a negative HIV serology and an undetectable viral load.
* Patient known to have one of the following concomitant genetic syndromes: Bloom syndrome, ataxia-telangiectasia, Fanconi anemia, Kostmann syndrome, Shwachman-Diamond syndrome or any other known bone marrow failure syndrome. Patients with Down syndrome are eligible for the study.
* Patients must not weigh < 17 kg.
* Patients must not have received prior therapy with a CD123 directed antibody or CD123 directed chimeric antigen receptor (CAR) T cells.
* Patients who have an uncontrolled infection are not eligible.
* Patients who have received a prior solid organ transplantation are not eligible.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.
* Known hypersensitivity to murine, yeast, or recombinant proteins; polysorbate 80; recombinant human serum albumin; benzyl alcohol; or any excipient contained in the flotetuzumab drug formulation. Additionally, those patients who have had a hypersensitivity reaction to etoposide that is considered likely related to polysorbate 80 are not eligible.
* Patients must refrain from driving a motor vehicle or operating heavy machinery while receiving flotetuzumab and for 30 days from the date of last study drug administration.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Lamble, Principal Investigator — Pediatric Early Phase Clinical Trial Network
Locations (19):
- United States (19):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Phase 1 Trial of the CD123 X CD3 DART Molecule Flotetuzumab (NSC#808294) in Children, Adolescents, and Young Adults with Relapsed or Refractory Acute Myeloid Leukemia.
Pre-assignment Details: Flotetuzumab for the Treatment of Pediatric Recurrent or Refractory Acute Myeloid Leukemia.
Groups:
- Part A Dose Level 1: 500 Nanograms/kg/Day; Part A Dose Level 2: 700 Nanograms/kg/Day: Patients receive flotetuzumab IV continuously for 28 days. Treatment repeats every 29 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive cytarabine intrathecally (IT) on days -6 to 0 prior to cycle 1. Patients may receive additional doses of cytarabine on day 1 of subsequent cycles per physician discretion.
Period: Overall Study
Arm/Group | Part A Dose Level 1: 500 Nanograms/kg/Day | Part A Dose Level 2: 700 Nanograms/kg/Day
Started | 7 | 9
Completed | 0 | 0
Not Completed | 7 | 9
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 3 | 7
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Dose Level 1: 500 Nanograms/kg/Day | Part A Dose Level 2: 700 Nanograms/kg/Day | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 8 | 15
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: Year] | 14 [3.0 to 17.0] | 15 [4.0 to 19.0] | 14.5 [3.0 to 19.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities Due to Flotetuzumab
Description: Number and percentage of patients experiencing dose limiting toxicities during cycle 1 that are possibly, probably, or definitely due to flotetuzumab by dose level and study part.
Time Frame: Up to 29 days
Population: Eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1: 500 Nanograms/kg/Day | Part A Dose Level 2: 700 Nanograms/kg/Day
Number analyzed (Participants) | 7 | 9
Participants | 1 | 1

2. Primary Outcome: Maximum Tolerated Dose or Recommended Phase 2 Dose of Flotetuzumab
Description: Estimated maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of Flotetuzumab defined by the maximum dose at which fewer than one-third of toxicity-evaluable participants experience a DLT. RP2D was established by study committee based off the toxicity profile of DL1 (500 ng/kg/day).
Time Frame: Up to 29 days
Population: Eligible patients
Measure: Number; unit: nanograms/kg/day
Groups:
- Treatment (Flotetuzumab, Cytarabine): Patients receive flotetuzumab IV continuously for 28 days. Treatment repeats every 29 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive cytarabine intrathecally (IT) on days -6 to 0 prior to cycle 1. Patients may receive additional doses of cytarabine on day 1 of subsequent cycles per physician discretion.
Arm/Group | Treatment (Flotetuzumab, Cytarabine)
Number analyzed (Participants) | 16
nanograms/kg/day | 500

3. Secondary Outcome: Maximum Concentration (C Max)
Description: Median with Minimum and Maximum for the maximum (peak) serum concentration measured on days 3-9 post-administration by dose level and study part.
Time Frame: Up to 9 days
Population: Eligible patients
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Part A Dose Level 1: 500 Nanograms/kg/Day | Part A Dose Level 2: 700 Nanograms/kg/Day
Number analyzed (Participants) | 6 | 8
pg/ml | 108.6 [0.0 to 139.6] | 147.6 [17.3 to 1835.4]

4. Secondary Outcome: Antitumor Activity of Flotetuzumab
Description: Number of response evaluable participants with response (CR/PR) using revised AML International Working Group criteria for response including CR: M1 bone marrow (<5% blasts), ANC at least 1000/mm3 and platelet count at least 100,000/mm3; CRp: platelet transfusion independence; CRi: without platelet transfusion independence, CRc: revision to normal karyotype; PR: decrease at least 50% in percentage of blasts to 5% to 25% in bone marrow aspirate.
Time Frame: Up to 2 years
Population: Response evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Part A Dose Level 1:500 Nanograms/kg/Day; Part A Dose Level 2: 700 Nanograms/kg/Day: Patients receive flotetuzumab IV continuously for 28 days. Treatment repeats every 29 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive cytarabine intrathecally (IT) on days -6 to 0 prior to cycle 1. Patients may receive additional doses of cytarabine on day 1 of subsequent cycles per physician discretion.
Arm/Group | Part A Dose Level 1:500 Nanograms/kg/Day | Part A Dose Level 2: 700 Nanograms/kg/Day
Number analyzed (Participants) | 7 | 8
Participants | 1 | 1

5. Other Pre Specified Outcome: Change in T-lymphocyte Population Numbers
Description: Changes in T cell number will be described and exploratory analysis will be conducted to assess their correlation with clinical features including occurrence of infections and response. Disease response will be assessed according to the revised acute myeloid leukemia (AML) International Working Group (IWG) criteria and will be reported descriptively. Analyses will be descriptive and exploratory and hypothesis-generating in nature.
Time Frame: Up to 180 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: CD123 Surface Expression
Description: CD123 expression will be analyzed in an exploratory fashion, both using a binary scale and using a continuous scale to evaluate whether there are correlations between CD123 expression and anti-leukemia effects. Analyses will be descriptive and exploratory and hypothesis-generating in nature.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 Years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Groups:
- Stratum 1 Dose Level 1: 500 nanograms/kg/day
- Stratum 1 Dose Level 2: 700 nanograms/kg/day
Arm/Group | Stratum 1 Dose Level 1 | Stratum 1 Dose Level 2
All-Cause Mortality (participants affected / at risk) | 0/7 | 2/9
Serious Adverse Events (participants affected / at risk) | 7/7 | 8/9
Other Adverse Events (participants affected / at risk) | 7/7 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1 Dose Level 1 (N=7) | Stratum 1 Dose Level 2 (N=9)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Alkalosis (Metabolism and nutrition disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 6 | 5
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 1
Cardiac disorders - Other, Decreased shortening fraction. (Cardiac disorders) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Creatinine increased (Investigations) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 2
Death NOS (General disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Fever (General disorders) | 0 | 2
Heart failure (Cardiac disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 2
Hypokalemia (Metabolism and nutrition disorders) | 4 | 5
Hypotension (Vascular disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
INR increased (Investigations) | 1 | 0
Infections and infestations - Other, VRE mastoiditis (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Lymphocyte count decreased (Investigations) | 6 | 6
Lymphocyte count increased (Investigations) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Nail infection (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 4 | 4
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Pericardial tamponade (Cardiac disorders) | 1 | 0
Platelet count decreased (Investigations) | 5 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Sepsis (Infections and infestations) | 2 | 2
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 1
Typhlitis (Gastrointestinal disorders) | 1 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
White blood cell decreased (Investigations) | 7 | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1 Dose Level 1 (N=7) | Stratum 1 Dose Level 2 (N=9)
Abdominal distension (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 2
Agitation (Psychiatric disorders) | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Aortic valve disease (Cardiac disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Blood bilirubin increased (Investigations) | 2 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 2 | 2
Capillary leak syndrome (Vascular disorders) | 2 | 4
Cardiac disorders - Other, Bigeminy PVCs (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, left ventricular trabeculations (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, mild dilation of left ventricle (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, mildly dilated left atrium (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, mildly elevated right ventricular systolic pressure (Cardiac disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chills (General disorders) | 3 | 1
Confusion (Psychiatric disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Creatinine increased (Investigations) | 1 | 3
Cushingoid (Endocrine disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 4 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 2
Dizziness (Nervous system disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Edema face (General disorders) | 2 | 2
Edema limbs (General disorders) | 2 | 3
Edema trunk (General disorders) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Eye pain (Eye disorders) | 1 | 0
Facial muscle weakness (Nervous system disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Fatigue (General disorders) | 4 | 4
Fever (General disorders) | 4 | 2
Fibrinogen decreased (Investigations) | 1 | 1
Flushing (Vascular disorders) | 2 | 2
GGT increased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 4 | 4
Heart failure (Cardiac disorders) | 1 | 0
Hematoma (Vascular disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 2
Hepatobiliary disorders - Other, "hepatomegaly with liver 3 cm below costal margin." (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disorders - Other, Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 1
Hepatobiliary disorders - Other, enlarged liver (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disorders - Other, hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 2
Hypertension (Vascular disorders) | 3 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 6
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 5
Hyponatremia (Metabolism and nutrition disorders) | 5 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 7
Hypotension (Vascular disorders) | 4 | 2
INR increased (Investigations) | 3 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Investigations - Other, C-reactive protein elevated (Investigations) | 0 | 1
Investigations - Other, C-reactive protein increased (Investigations) | 1 | 0
Investigations - Other, CRP increased (Investigations) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 1
Lethargy (Nervous system disorders) | 1 | 1
Localized edema (General disorders) | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 1
Lymphocyte count increased (Investigations) | 1 | 2
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Mitral valve disease (Cardiac disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 5 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Nervous system disorders - Other, "waxing/waning mental status despite holding sedating meds." (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, changes in visual perception (Nervous system disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Pain (General disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 2 | 1
Pericardial effusion (Cardiac disorders) | 2 | 2
Periorbital edema (Eye disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1
Phlebitis infective (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Proteinuria (Renal and urinary disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary valve disease (Cardiac disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3
Renal and urinary disorders - Other, Nephromegaly (Renal and urinary disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — "New retrocardiac opacity, may reflect atelectasis and/or infection. New somewhat patchy opacity porjecting over the medial right lower lung zone, which may reflect infection and/or atelectasis
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — diminished breath sounds: bases and tachypnic." Progress Note 02/04/20 08. "work of breathing and abdominal competition
Respiratory, thoracic and mediastinal disorders - Other, Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, Tachypnea noted... no respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, bradypnea during sleep (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, left hemidiaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 5 | 6
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0 — Ecchymosis: distributed throughout upper and lower extremities
Skin and subcutaneous tissue disorders - Other, "spot of petechia to right thigh." (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, Clammy (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, Erythematous rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, Presumed GT cellulutus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, abdominal skin nodules (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, erythema (intermittent) (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, ingrown toenail (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0 — Scattered petechiae to forehead and around eyes bilaterally.
Skin infection (Infections and infestations) | 1 | 0
Somnolence (Nervous system disorders) | 2 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Stomach pain (Gastrointestinal disorders) | 2 | 0
Surgical and medical procedures - Other, Surgical and Medical Procedure (Surgical and medical procedures) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urine discoloration (Renal and urinary disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 6
Weight gain (Investigations) | 5 | 1
Weight loss (Investigations) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT04158739/Prot_SAP_001.pdf
  • Informed Consent Form (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT04158739/ICF_000.pdf